CLINICAL TRIAL: NCT06439095
Title: Evaluation of IL-2, IL-5 and IL-17 Expression Levels in Saliva of Patients Treated With Stainless Steel Crowns
Brief Title: Interleukin-2 (IL-2), Interleukin-5 (IL-5) and Interleukin-17 (IL-17) Levels of Patients With Stainless Steel Crowns
Status: Completed | Type: Observational
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Burçin AVCI, Assistant Professor, Yuzuncu Yil University
Other Study IDs: YYU-BAVCI-01
Record Dates: First submitted 2024-05-27; First posted 2024-06-03 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Saliva; Dental Crown; Nickel Sensitivity
Keywords: Saliva; Dental crown; Gene expression
MeSH Terms: interventions — Hydrogen-Ion Concentration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva of patients using stainless steel crown
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stainless Steel Crown Group: Participants in this group received stainless steel crowns on posterior teeth. Salivary samples were collected before treatment (pre-treatment) and 7 days after treatment. IL-2, IL-5, and IL-17 gene expression levels were measured using Real-Time PCR. Additionally, salivary pH and the concentration of nickel, chrome ions were analyzed using atomic absorption spectrophotometry.
  Interventions: Genetic: Salivary Collection; Diagnostic Test: Ph and ion level measurement of saliva

INTERVENTIONS:
Genetic: Salivary Collection — Expression levels of IL-2, IL-5 and IL-17 in the saliva of individuals aged 3-9 years who underwent stainless steel crown will be recorded before and after the procedure. Before the saliva sample collection procedure, the patient will be asked to rinse their mouth with sterile water and then spit into sterile plastic cups. After collecting approximately 3 ml of saliva, the saliva will be transferred to appropriate eppendorfs and stored at -40 degrees Celsius. For the second post-procedure, the same algorithms will be applied for saliva collection seven days after the crown procedure.
Diagnostic Test: Ph and ion level measurement of saliva — Salivary concentration of nickel, chrome ions will be measured using an atomic absorption spectrophotometer.

SUMMARY:
The aim of this study is to investigate whether nickel hypersensitivity following stainless steel crown treatment in children aged 3-9 leads to an increase in IL-2, IL-5, and IL-17 levels by analyzing saliva samples. By doing so, the study seeks to prevent potential hypersensitivity reactions after stainless steel crown treatment.

The main question it aims to answer is:

Which interleukin level increases in the controls 1 week after stainless steel crowns are applied? Researchers will investigate whether there is a significant increase in interleukin levels in children's saliva before and after the procedure.

Participants will:

They will provide saliva samples before stainless steel crowns are applied They will visit the clinic after 1 week for check-ups and tests.

DETAILED DESCRIPTION:
Expression levels of IL-2, IL-5 and IL-17 in the saliva of individuals aged 3-9 years who underwent stainless steel crown will be recorded before and after the procedure. Before the saliva sample collection procedure, the patient will be asked to rinse their mouth with sterile water and then spit into sterile plastic cups. After collecting approximately 5 ml of saliva, the saliva will be transferred to appropriate eppendorfs and stored at -40 degrees Celsius. For the second post-procedure, the same algorithms will be applied for saliva collection seven days after the crown procedure. Also ph value and ion levels of saliva will be measured.

ELIGIBILITY:
**Inclusion Criteria:**

* Patients with teeth requiring stainless steel crowns due to having caries on two or more surfaces.
* Pediatric patients between 3-9 years old

**Exclusion Criteria:**

* Patients having any dental materials, such as fillings, fissure sealants, root canal treatments, or space maintainers
* Patients with known allergies to various foods and materials.
* Patients with systemic diseases that affect the immune system.
* Patients with a history of chemotherapy or radiotherapy.

Ages: 3 Years to 9 Years | Sex: All
Age Groups: Child
Study Population: The patients living in Van city
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Burçin Avcı, DDS, MSc, Principal Investigator — Yuzuncu Yil University
Locations (1):
- Yüzüncü Yil University, Van, Tuşba, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Avci B, Koc A, Kaya S. Evaluation of Salivary IL-2, IL-5, and IL-17 Levels in Paediatric Patients Treated With Stainless Steel Crowns. Int J Paediatr Dent. 2025 Dec 30. doi: 10.1111/ipd.70071. Online ahead of print. PMID 41469209

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from pediatric dental clinics and selected based on the need for stainless steel crown placement.
Pre-assignment Details: Twelve patients were enrolled according to the study protocol and all twelve commenced the study.
Groups:
- Stainless Steel Crown Group: Patients received stainless steel crowns, and salivary IL-2, IL-5, and IL-17 gene expression levels were measured at baseline and after 7 days.
Period: Overall Study
Arm/Group | Stainless Steel Crown Group
Started | 12
Completed | 10
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Baseline data was collected from all 12 participants before 2 participants were withdrawn due to loss to follow-up.
Arm/Group | Stainless Steel Crown Group
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 6.4 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Baseline IL-2, IL-5, and IL-17 Expression Status [Mean (Standard Deviation); unit: Relative Expression Units] — Average baseline IL-2, IL-5, and IL-17 expression levels measured in saliva before SSC procedure.
  Relative Expression Units
    Baseline IL-2 Expression (Relative Units) | 1.0 (0.1)
    Baseline IL-5 Expression (Relative Units) | 1.0 (0.15)
    Baseline IL-17 Expression (Relative Units) | 1.0 (0.2)

OUTCOME MEASURES:

1. Primary Outcome: IL-2, IL-5, IL-17 Expression Level (Fold Change)
Description: Relative gene expression analysis was performed using quantitative PCR (qPCR) with appropriate primers. The results were reported as fold change relative to baseline values.
Time Frame: Sample collection at baseline (Day 0) and 7 days after treatment
Population: Of 12 enrolled participants, data from 10 participants were included in the final analysis due to complete sample availability.
Measure: Mean (Standard Deviation); unit: Fold Change
Groups:
- Stainless Steel Crown Group: Patients received stainless steel crowns on posterior teeth. Salivary IL-2, IL-5, and IL-17 gene expression levels were measured before treatment and 7 days after.
Arm/Group | Stainless Steel Crown Group
Number analyzed (Participants) | 10
Fold Change
  Day 7 IL-2 Expression (Fold Change) | 1.2 (0.4)
  Day 7 IL-5 Expression (Fold Change) | 1.8 (0.3)
  Day 7 IL-17 Expression (Fold Change) | 4.5 (1.7)

ADVERSE EVENTS:
Time Frame: Baseline until 7 days post-treatment
Description: Adverse events were monitored through systematic clinical examination and parental interviews.
Arm/Group | Stainless Steel Crown Group
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
The small sample size and short 7-day follow-up limit the generalizability and long-term interpretation of the results. The before-and-after design reduces variability but does not fully control for genetic, immune, or environmental factors. Larger randomized studies are needed to confirm these findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT06439095/Prot_SAP_ICF_000.pdf